CLINICAL TRIAL: NCT00450229
Title: Phase Ib Placebo-Controlled Trial of Diindolylmethane (BR-DIM) in the Study of the Modulation of Intermediate Endpoint Markers in Patients With Prostate Cancer Who Are Undergoing Prostatectomy
Brief Title: Diindolylmethane in Treating Patients Undergoing Surgery for Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2009-00905; CO05816; CDR0000656281; H2006-0255; N01CN35153 (NIH)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-05

CONDITIONS: Adenocarcinoma of the Prostate; Prostate Cancer; Stage I Prostate Cancer; Stage II Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3,3'-diindolylmethane

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm I (Experimental): Patients receive low-dose, nutritional-grade oral diindolylmethane (DIM) twice daily for 21-28 days in the absence of disease progression or unacceptable toxicity. Treatment may continue for up to 60 days, if surgery is delayed.
  Interventions: Drug: diindolylmethane; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (Experimental): Patients receive high-dose, nutritional-grade oral DIM twice daily as in arm I.
  Interventions: Drug: diindolylmethane; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm III (Placebo Comparator): Patients receive oral placebo twice daily for 21-28 days in the absence of disease progression or unacceptable toxicity. Treatment may continue for up to 60 days, if surgery is delayed.
  Interventions: Drug: placebo; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: diindolylmethane — Given PO
  Other Names: DIM
  Arms: Arm I; Arm II
Drug: placebo — Given PO
  Other Names: PLCB
  Arms: Arm III
Procedure: therapeutic conventional surgery — Undergo surgical resection
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Giving diindolylmethane, a substance found in cruciferous vegetables, may help doctors learn more about how diindolylmethane is used by the body. This randomized phase I trial is studying the side effects and best dose of diindolylmethane compared with a placebo in treating patients undergoing radical prostatectomy for stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare neoadjuvant prostatic diindolylmethane (DIM^) concentrations in patients with stage I or II adenocarcinoma of the prostate treated with DIM vs placebo prior to radical prostatectomy.

SECONDARY OBJECTIVES:

I. Compare the ratio of urinary 2-hydroxyestrone:16-hydroxyestrone in patients treated with these regimens.

II. Compare plasma levels of total prostate-specific antigen (PSA) in patients treated with these regimens.

III. Compare serum testosterone levels in patients treated with these regimens. IV. Compare the ratio of plasma insulin-like growth factor (IGF)-1:IGF binding protein-3 in patients treated with these regimens.

V. Compare cytochrome p450 mRNA expression of CYP1A1, CYP1A2, CYP2B1, and CYP3A enzymes in circulating polymorphonuclear leukocytes (PMNs) and in fresh frozen tissue in patients treated with these regimens.

VI. Compare DIM blood steady-state concentrations in patients treated with these regimens.

VII. Identify polymorphisms of CYP1A1, CYP1A2, CYP2B1, and CYP3A in circulating PMNs in patients treated with these regimens.

VIII. Compare tissue levels of PSA, androgen receptor, Ki-67, and caspase 3 in patients treated with these regimens.

OUTLINE:

This is a randomized, placebo-controlled, multicenter study. Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive low-dose, nutritional-grade oral diindolylmethane (DIM) twice daily for 21-28 days in the absence of disease progression or unacceptable toxicity. Treatment may continue for up to 60 days, if surgery is delayed.

Arm II: Patients receive high-dose, nutritional-grade oral DIM twice daily as in arm I.

Arm III: Patients receive oral placebo twice daily for 21-28 days in the absence of disease progression or unacceptable toxicity. Treatment may continue for up to 60 days, if surgery is delayed.

Patients in all arms undergo surgical resection of their tumor within 1 day after completion of DIM or placebo.

Patients undergo blood, tissue, and urine sample collection periodically during study for immunohistochemical (IHC)/molecular analyses and pharmacokinetic and pharmacogenomic correlative studies. Patient specimens are assessed for DIM levels in plasma and tissue (by liquid chromatography/mass spectrometry [LC/MS]) and for biologic response to DIM (by TUNEL assay). Intermediate biomarkers of DIM activity are also assessed, including urinary 2-hydroxyestrone:16-hydroxyestrone ratio (by LC/MS assay), plasma total prostate-specific antigen (PSA), plasma insulin-like growth factor (IGF)-1:IGF binding protein-3 ratio (by ELISA), and tissue androgen receptor, PSA, Ki-67, and caspase 3 (by immunohistochemistry). Cytochrome p450 induction and gene expression (CYP1A1, CYP1A2, CYP2B1, CYP3A) are also assessed in tissue and plasma by semiquantitative real-time polymerase chain reaction.

ELIGIBILITY:
Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Clinical stage T1 or T2 a, b, or c (stage I-II disease)
* Disease is confined within the prostate gland
* Candidate for radical prostatectomy
* ECOG performance status (PS) 0-1 OR Karnofsky PS 80-100%
* WBC normal
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* AST =< 1.5 times upper limit of normal
* Creatinine =< 2.0 mg/dL
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to diindolylmethane (DIM^), any of the inactive ingredients contained in BioResponse-DIM^NG or placebo, or to compounds of similar chemical or biologic composition
* No concurrent uncontrolled illness including, but not limited to, any of the following: Ongoing or active infection, Symptomatic congestive heart failure, Unstable angina pectoris, Cardiac arrhythmia, No psychiatric illness or social situation that would preclude study compliance
* No prior chemotherapy, hormonal therapy, brachytherapy, or external radiotherapy for prostate cancer
* No concurrent nonsteroidal anti-inflammatory drugs, including acetylsalicylic acid, ibuprofen, naproxen sodium, or cyclooxygenase-2 inhibitors
* No concurrent systemic therapy for any other cancer
* No other concurrent investigational agents
* No concurrent p450 inducers or inhibitors, including any of the following: Carbamazepine, Clarithromycin, Fluconazole, Fosphenytoin, Itraconazole, Ketoconazole, Phenobarbital, Phenytoin, Rifabutin, Rifampin
* No concurrent finasteride or dutasteride
* No more than 1 serving of cruciferous vegetables per day for duration of study
* Cruciferous vegetables include the following: broccoli, cauliflower, brussels sprouts, cabbage, arugula, watercress, bok-choy, turnip greens, mustard greens, collard greens, rutabaga, Napa or Chinese cabbage, radishes, turnips, kohlrabi, and kale
* Bilirubin normal
* At least 21 days since prior surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Tissue levels of DIM | Up to 5 years
  The distribution of levels of DIM will be summarized by treatment arm with descriptive statistics. For the primary comparison between the placebo group and the DIM groups combined, tissue levels of DIM will be compared using Student t-test. In the case of violation of normality assumptions, an appropriate transformation of the data such as logarithm will be considered or a nonparametric test such as Wilcoxon rank-sum test will be used for comparison. A dose-response relation will be explored based on the analysis of covariance (ANCOVA).

SECONDARY OUTCOMES:
Urinary 2-hydroxyestrone/16-hydroxyestrone ratio | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
Total PSA | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
Serum testosterone | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
IGF1:IGFBP-3 ratio | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
Tissue measures of messenger RNA of CYPs (CYP1A2, CYP1A1, CYP2B1, CYP3A) | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
DIM blood steady-state concentrations | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.
Measures of androgen receptor, PSA, Ki-67, caspase 3, and TUNEL | Up to 5 years
  Will be summarized by treatment arm with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gee, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States